CLINICAL TRIAL: NCT00581152
Title: The Role of TBX3 in Human ES Cell Differentiation
Status: Withdrawn | Type: Observational
Why Stopped: IRB suspension
Sponsor: University of California, Irvine (Other)
Collaborators: CIRM SEED Grant (Unknown)
Responsible Party: Sponsor
Other Study IDs: OCRT07015 [HS# 2007-5848]; HS# 2007-5848
Record Dates: First submitted 2007-12-18; First posted 2007-12-27 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: TBX3; Cell Differentiation
Keywords: TBX3

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — NIH-approved cell lines will be available at the Sue and Bill Gross Stem Cell Research Core Facility at the University of California, Irvine. Non-NIH-approved cell lines will be obtained from Sue & Bill Gross Stem Cell Core at UC Irvine.
Oversight: Data Monitoring Committee: No

SUMMARY:
Stem cells can develop into every cell, every tissue and every organ in the human body, e.g., they can make any kind of cells in the human body. Stem cells reproduce themselves many times over and over. Their almost limitless potential has made stem cells a significant focus of medical research. But before scientists can use stem cells for medical purposes, they must first learn how to harness their power. They cannot treat disease until they learn how to manipulate stem cells to get them to develop into specific tissues or organs.

We know that turning genes on and off is crucial to the process differentiation, so we can add some factor into the culture dish and observe stem cells to differentiate into specific types of cells. But some sort of signal is needed to actually trigger the stem cells to differentiate. We are still searching for that signal. If we can ultimately learn how to direct stem cells to differentiate into one type of tissue or another, then we can use them to treat patients. In this proposal, we will first examine this step.

We propose a novel approach to understanding differentiation of human embryo stem (hES) cells, by studying TBX3, a protein called a transcription factor that controls the expression of other genes. In humans, the loss of function of TBX3 causes Ulnar-Mammary Syndrome, a genetic disorder that can pass from one generation to the next. Furthermore, our preliminary results show that TBX3 is downstream mediator of another protein, BMP4. BMP4 is a known key regulator for hES cell differentiation. Thus, TBX3 is an attractive candidate as a downstream mediator of BMP4 in hES cell differentiation. We will test TBX3 effects on hES cell differentiation if down-regulate TBX3 in hES cells with a technology called siRNA knockdown. We will identify the genes controlled by TBX3 with a recently invented powerful technology called CHIP-GLAS. This technique allows us to examine thousands of genes on a small chip in a single experiment. We expect that the innovative experiments proposed here will open a new avenue to understanding the signal of hES cell differentiation.

DETAILED DESCRIPTION:
PURPOSE OF STUDY The purpose of this study is to understand what triggers stem cells to differentiate into one type of tissue or another. The study of TBX3, a protein called a transcription factor that controls the expression of other genes, shows that it is a downstream mediator of the protein BMP4, a known key regulator for hES cell differentiation.

Hypothesis and Aims

To understand the role of TBX3 in hES cell differentiation, we hypothesize that TBX3 is a downstream mediator of BMP4 and play an important role in hES cell differentiation. We propose the following specific aims:

1. To examine TBX3 function in hES cell differentiation. NIH approved hES cells will be cultured in a conditioned medium with BMP4 to induce differentiation and TBX3 expression. TBX3 will be knocked down with siRNA technology. The cell morphology and biochemical changes will be examined for the effects of TBX3 knockdown on hES cell differentiation, including testing human ß-CG estradiol and progesterone. The gene expression profile will also be examined with Affymetrix gene expression chip and verified with real-time RT-PCR.
2. To identify the genome-wide downstream targets directly bound by TBX3 in hESC with Chromatin immunoprecipitation-guided ligation and selection (CHIP-GLAS). To identify the targets of TBX3 in BMP4-induced hES cells, we will perform ChIP-GLAS analysis. CHIP-GLAS is a novel high-throughput technique with combination of chromatin precipitation and oligonucleotide-based microarray. This technology will allow us to identify the genome-wide downstream target genes directly bound by TBX3 in hES cells.

We expect that the proposed experiments will identify a key regulator for hES cell differentiation and open a new avenue to understanding the function of TBX3 in hES cells. The CHIP-GLAS promoter array provides us a cutting edge tool and allows us to examine the broad function of TBX3. We anticipate that the study will significantly enhance our understanding of TBX3 function in hES cell differentiation.

STUDY DESIGN NIH-approved cell lines will be available at the Sue and Bill Gross Stem Cell Research Core Facility at the University of California, Irvine. Non-NIH-approved cell lines will be obtained from Sue & Bill Gross Stem Cell Core at UC Irvine.

Environment: Huang Lab is currently supported by the Helen and Larry Hoag Foundation and the Susan Komen Foundation. There are no active grants from the federal government. Previously, Dr. Huang was supported by K23 and R03 grants. They were completed in 2004 and 2006, respectively. No equipment was purchased with the funds from the federal grants. As all equipment currently in Huang lab was purchased with the UCI startup fund or with private funds, there is no conflict with government regulations.

At University California, Irvine, Sue and Bill Gross Stem Cell Research Center will be a key component of the Stem Cell Core Facility. This facility provides stem cell technology and resources to the UCI faculty (Please see attached letter). By merging technical and scientific expertise in a number of essential disciplines, the Core harbors a diverse tool kit for the exploration of multiple aspects of stem cell biology. The Core also provides a knowledge base for differentiating, genetically modifying and assaying human embryonic stem cells (hESCs) in support of multiple stem cell projects on campus and in the surrounding area. All services and procedures are performed in accordance with good quality assurance and record keeping practices pursuant to standard operating procedures and good laboratory practices.

The Sue and Bill Gross Stem Cell Research Center The human embryonic stem (hES) cell core facility of the Sue and Bill Gross Stem Cell Research Center opened in April 2006. It occupies approximately 10,000 square feet of space in the research park immediately adjacent to the University of California, Irvine campus. Approximately $1.7 million were committed by the UCI to fully equip the facility for all aspects on hES cell research. Further gifts totaling $236,687 from the Fuji Foundation and the Nichols Foundation provided additional major equipment and supplies that are available for all investigators. The facility was set up as a Federal-free zone in which investigators can to carry out all aspects of hES cell research. Individual rooms are equipped with tissue culture biosafety cabinets, CO2 incubators, an inverted microscope, a dissecting microscope, digital imaging equipment, a centrifuge, a water bath and a dedicated refrigerator and freezer. Ten such tissue culture set-ups as well as standard lab bench space are available to UCI investigators and visitors.

The facility also has major pieces of equipment needed for hES cell analysis such as a Zeiss 510 Meta Two-Photon Confocal Microscope. The facility will shortly have a BD LSR II Flow cytometer and a BD FacsAria cell sorter. Pretested reagents will be available to investigators through the core facility. These will include medium components, growth factors, feeder cells, gelatin, Matrigel, antibodies and primers to assay stem cell marker expression. In addition, the core facility will assist in karyotype analysis and tumor formation tests of hES cells.

ELIGIBILITY:
Inclusion Criteria:

* none

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: No subjects will be consented for this study. Approximately 2 to 4 cell lines will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2010-08-28 (Actual); Study Completion 2010-08-28 (Actual)

PRIMARY OUTCOMES:
The cell morphology and biochemical changes will be examined for the effects of TBX3 knockdown on hES cell differentiation, including testing human ß-CG estradiol and progesterone. | 3 years
To identify the targets of TBX3 in BMP4-induced hES cells, we will perform ChIP-GLAS analysis. CHIP-GLAS will allow us to identify the genome-wide downstream target genes directly bound by TBX3 in hES cells. | 3 years